CLINICAL TRIAL: NCT03423277
Title: Easy Stretch Toolkit: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-0005
Record Dates: First submitted 2018-01-16; First posted 2018-02-06 (Actual); Results first posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Facial Injuries
MeSH Terms: conditions — Facial Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Easy Stretch Toolkit (Experimental): All participants will be using one or more of devices for 60 minutes 2 times per day for the duration of the 8 week trial. Prescriptive instructions for specific intraoral placements will be given based on the participant's deficit areas.
  Interventions: Device: Easy Stretch Toolkit

INTERVENTIONS:
Device: Easy Stretch Toolkit — Study the use of novel intraoral tools for management of facial burns and other facial disorders

SUMMARY:
To research the use of a novel set of intraoral tools called the Easy Stretch Toolkit for the therapeutic management of facial burns and other facial disorders.

DETAILED DESCRIPTION:
In this initial pilot study, we plan to recruit 20 adult or pediatric patients who have sustained facial burns or who have sustained a facial injury resulting in scarring, tightness, limited range of motion of facial skin or musculature, or fibrosis to complete the 8 week treatment. Participants will need to be able to attend a weekly telehealth or in person session with the investigators and complete the entire 8 week prescriptive program. Participants will be outpatient. A facial injury can be any disorder that results in scarring, tightness, limited range of motion of facial skin or musculature or fibrosis. Facial burn injury or facial injury is defined as an injury to the midface or lower half of the face and may be unilateral or bilateral. Participants must be in the chronic phase of recovery. Chronic burns are defined as those burns that are not in the acute healing phase, ie., there are no concerns for injury to new or healing skin or wound dehiscence.

ELIGIBILITY:
Inclusion criteria:

1. Age 7-80
2. Male or Female Sex
3. Patients who have sustained a facial burn and are now in the chronic phase, or any patient experiencing facial tightness or limited range of motion due to other problems, including patients s/p radiation to the head and neck, trauma, scarring and scleroderma
4. Chief complaint(s) of limited mouth opening, difficulty chewing or speaking, decreased range of motion for oral structures, and/or limited facial expressions
5. Subject or caregiver (parent or guardian, in case of pediatric population) must be able to give informed consent
6. Subject or caregiver (parent or guardian, in case of pediatric population) must be able to perform exercises at home and must be able to record time spent using the devices.
7. Participants who are undergoing other treatment methods such as use of compression garments, skin grafting, radiation or other facial surgery, etc must suspend all of these treatments for the duration of the 2 month trial.
8. Internet access including access to FaceTime, Skype or Zoom and email access if electing telehealth option for enrollment

Exclusion criteria:

1. planned or unplanned surgeries for facial skin grafting around lips or nose or oral commissure release during the upcoming 8 weeks
2. completion of any massaging or other stretching exercises or programs not specified by the investigators
3. use of new creams or topical treatments for the duration of enrollment in the study.
4. acutely burn-injured patients
5. incarceration, or pregnancy

Ages: 7 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-02-28 (Actual); Primary Completion 2022-11-07 (Actual); Study Completion 2022-11-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lori Arguello, Principal Investigator — employee of University of Texas Medical Branch; Kathleen Kerr, Study Director — employee of University of Texas Medical Branch
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Clayton NA, Ward EC, Maitz PK. Orofacial contracture management outcomes following partial thickness facial burns. Burns. 2015 Sep;41(6):1291-7. doi: 10.1016/j.burns.2015.02.015. Epub 2015 Jun 26. PMID 26120089
- [Background] Clayton NA, Ward EC, Maitz PK. Intensive swallowing and orofacial contracture rehabilitation after severe burn: A pilot study and literature review. Burns. 2017 Feb;43(1):e7-e17. doi: 10.1016/j.burns.2016.07.006. Epub 2016 Aug 26. PMID 27575671
- [Background] Macintyre L, Baird M. Pressure garments for use in the treatment of hypertrophic scars--a review of the problems associated with their use. Burns. 2006 Feb;32(1):10-5. doi: 10.1016/j.burns.2004.06.018. PMID 16413399
- [Background] Atiyeh BS, El Khatib AM, Dibo SA. Pressure garment therapy (PGT) of burn scars: evidence-based efficacy. Ann Burns Fire Disasters. 2013 Dec 31;26(4):205-12. PMID 24799851
- [Background] Clayton NA, Ellul G, Ward EC, Scott A, Maitz PK. Orofacial Contracture Management: Current Patterns of Clinical Practice in Australian and New Zealand Adult Burn Units. J Burn Care Res. 2017 Jan/Feb;38(1):e204-e211. doi: 10.1097/BCR.0000000000000351. PMID 27359188
- [Background] Parry I, Sen S, Palmieri T, Greenhalgh D. Nonsurgical scar management of the face: does early versus late intervention affect outcome? J Burn Care Res. 2013 Sep-Oct;34(5):569-75. doi: 10.1097/BCR.0b013e318278906d. PMID 23816994
- [Background] Hadlock TA, Urban LS. Toward a universal, automated facial measurement tool in facial reanimation. Arch Facial Plast Surg. 2012 Jul-Aug;14(4):277-82. doi: 10.1001/archfacial.2012.111. PMID 22508895
- [Background] Marur T, Tuna Y, Demirci S. Facial anatomy. Clin Dermatol. 2014 Jan-Feb;32(1):14-23. doi: 10.1016/j.clindermatol.2013.05.022. PMID 24314374
- [Background] Jorge JJ Jr, Pialarissi PR, Borges GC, Squella SA, de Gouveia Mde F, Saragiotto JC Jr, Goncalves VR. Objective computerized evaluation of normal patterns of facial muscles contraction. Braz J Otorhinolaryngol. 2012 Apr;78(2):41-51. doi: 10.1590/S1808-86942012000200008. PMID 22499369
- [Background] Feng G, Zhuang Y, Gao Z. Measurement and analysis of associated mimic muscle movements. J Otol. 2015 Mar;10(1):39-45. doi: 10.1016/j.joto.2015.06.001. Epub 2015 Aug 1. PMID 29937780
- [Background] Coulson SE, Croxson GR, Gilleard WL. Quantification of the three-dimensional displacement of normal facial movement. Ann Otol Rhinol Laryngol. 2000 May;109(5):478-83. doi: 10.1177/000348940010900507. PMID 10823477
- [Background] VanSwearingen JM, Brach JS. The Facial Disability Index: reliability and validity of a disability assessment instrument for disorders of the facial neuromuscular system. Phys Ther. 1996 Dec;76(12):1288-98; discussion 1298-300. doi: 10.1093/ptj/76.12.1288. PMID 8959998

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Easy Stretch Toolkit
Started | 8
Completed | 4
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Easy Stretch Toolkit
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 6
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Change in the Facial Range of Motion at Baseline and Week 8
Description: Facial measurements taken during select facial movements/expressions assessed by software program created at UTMB specifically for this project. The degree of change in facial movements will be assessed with 9 facial postures (face at rest, nose wrinkle, gentle smile, broad smile with lips closed, broad smile with teeth together, voice "eee", voice "ooo", pucker lips and open mouth wide), which will be photographed weekly. Two examples of the facial landmarks to be plotted and measured during each of the above expressions include right pupil to outside of right nare and length of philtrum, with the goal of measuring change over time with use of the Easy Stretch devices. Each of these measurements will produce a length in millimeters. Cumulative average of measurements will be reported per facial posture per participant.
Time Frame: 8 weeks
Population: 8 enrolled, only 4 completed program
Measure: Median (Full Range); unit: mm
Groups:
- Facial Measurement Data: Facial measurement data were collected at week 1 and week 8 for each participant as distance between 2 facial landmarks as the participant completed requested facial expressions such as "open mouth wide" and "gentle smile". Data was collected for 13 measurements across 9 facial expressions.
Arm/Group | Facial Measurement Data
Number analyzed (Participants) | 4
mm
  At Rest | -16.12 [-20.56 to 7.99]
  Wrinkle Nose | -.08 [-16.77 to 6.43]
  Gentle Smile | -7.34 [-18.78 to 3.02]
  Broad Smile Lips Closed | 4.47 [-10.89 to 16.47]
  Broad Smile Show Teeth | -3.77 [-13.55 to 11.30]
  Say 'ooo' | 0.53 [-11.24 to 12.03]
  Say 'eee' | -1.86 [-6.68 to 12.173]
  Pucker | -2.97 [-12.66 to 14.84]
  Open Your Mouth Wide | 0.14 [-13.95 to 8.57]

2. Secondary Outcome: Change in the Facial Disability Index Scores From Baseline to Week 8
Description: The Facial Disability Index (FDI) is a validated quality-of-life questionnaire consisting of 10 items, each scored on a 0-5 scale. Five items assess physical function and five items assess social well-being and function. Raw subscale scores are transformed according to standard FDI scoring procedures to yield physical function scores ranging from 0 to 100 and social function scores ranging from 0 to 100.
  The total Facial Disability Index score is calculated by summing the transformed physical and social subscale scores, resulting in a total score range of 0 to 200. Higher scores indicate better facial function and quality of life, while lower scores indicate greater facial disability.
Time Frame: baseline and week 8
Measure: Mean (Full Range); unit: score on a scale
Groups:
- Facial Disability Index Score: The Facial Disability Index is the name of a quality-of-life questionnaire that will be used for this study. It consists of 10 questions, with a scale of 0-5 for each question. 5 questions relate to physical function, and 5 questions relate to social well-being and function. The combined score provides an overall facial disability index score. A higher is a better outcome.
Arm/Group | Facial Disability Index Score
Number analyzed (Participants) | 4
score on a scale
  baseline | 129.5 [78 to 170]
  8 weeks | 151.5 [105 to 183]

ADVERSE EVENTS:
Time Frame: 8 weeks for each participant or the duration that they were enrolled in the study
Description: reviewed with each participant at the start of each session to ensure no adverse events had occurred during the use of the tools
Groups:
- Easy Stretch Toolkit: All participants will be using one or more of devices for 60 minutes 2 times per day for the duration of the 8-week trial. Prescriptive instructions for specific intraoral placements will be given based on the participant's deficit areas.
  Easy Stretch Toolkit: Study the use of novel intraoral tools for management of facial burns and other facial disorders.
Arm/Group | Easy Stretch Toolkit
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-01): https://cdn.clinicaltrials.gov/large-docs/77/NCT03423277/Prot_SAP_000.pdf